CLINICAL TRIAL: NCT03584594
Title: Prepepsin, the Improvement of the Early Inflammatory Biomarkers Strategy for the Diagnostics of Sepsis in Critically Ill Patients
Brief Title: Presepsin in the Diagnosis of Sepsis in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: Public Health Institute Ostrava (Unknown)
Responsible Party: Sponsor
Other Study IDs: KARIM-08-PSEPOVA
Record Dates: First submitted 2018-06-15; First posted 2018-07-12 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Sepsis; Infection
Keywords: presepsin; biomarkers; sepsis; diagnosis
MeSH Terms: conditions — Sepsis; Infections; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Residual blood samples remaining after performing all necessary standard and indicated blood examinations and analyses will be used to determine the level of presepsin, as the potential new biomarker of sepsis in critically ill patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Presepsin assessment: Residual blood samples after performing all necessary blood examinations and analyses will be used to determine the level of presepsin, as the potential new biomarker of infection.
  Interventions: Diagnostic Test: Presepsin measurement

INTERVENTIONS:
Diagnostic Test: Presepsin measurement — Presepsin measurements are performed with PathFast immunoassay analytical system on the ICU, bedside method. (Mitsubishi Chemical, Japan).

SUMMARY:
Sepsis is one of the most common causes of death worldwide. It is caused by a complex of inadequate host responses to infection. Sepsis remains a major challenge of modern intensive care medicine. Despite recent improvements, the incidence of sepsis in critically ill patients increases steadily (25%) and mortality rates remain unacceptably high (30%). It is difficult to distinguish the sepsis from the non-infectious systemic inflammatory response syndrome. Early identification of the origin of infection can help dramatically to improve outcome and reduce mortality. That is why clinicians need fast, reliable and specific biomarkers for sepsis recognition.

DETAILED DESCRIPTION:
Comparison between the detection of novel early inflammatory biomarker (PSEP) and the others normally used biomarkers (c-reactive protein - CRP, interleukin 6 - IL6, procalcitonin - PCT) in the early diagnosing of sepsis in the critically ill patients A broad range of clinical and laboratory parameters are combined (Surviving sepsis campaign, international guidelines) for early sepsis identification: white blood cells (WBC), C-reactive protein (CRP), interleukin 6 (IL-6), procalcitonin (PCT).

An ideal biomarker should be a fast and specific increase in sepsis, short half-life, rapid decrease after administration of an effective therapy and fast (bed-side) method of determination. None of the current biomarkers have all of these characteristics.

We investigate the diagnostic accuracy of presepsin compared to other biomarkers (WBC, PCT, IL6, CRP) for infection or sepsis, defined according to Sepsis-3 definition (Singer, JAMA 2016) in adult patients admitted to ICU with suspected sepsis.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* diagnosis of sepsis from qSOFA (quick Subsequent Organ Failures Assessment)
* need of vasopressors for mean arterial pressure (MAP) ≥ 65 mmHg
* lactate levels ≥ 2mmol/l despite adequate volume resuscitation

Exclusion Criteria:

* age below 18 years
* terminal state of disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a minimum 18 years admitted to ICU (surgical, traumatic, medical patients), who had proven criteria for sepsis, septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Serum concentration of Presepsin | 47 months
  Serum concentration of Presepsin in patients with sepsis or septic shock will be compared to PCT, IL6 and CRP results.
Area under the Receiver-operating characteristic Curve | 47 months
  Area under the Receiver-operating characteristic Curve (ROC-AUC) of the presepsin and other biomarkers (PCT, IL6, CRP) for diagnostic value of any biomarker will be analysed on a scale 0-100.

SECONDARY OUTCOMES:
Correlation of serum concentration of presepsin with detection of microbial agents | 47 months
  Comparison of presepsin concentration in serum with the results of culture/microscopy of a pathogen from a clinical focus using methods of classical microbiology. In patients with risk factors for invasive mycosis, comparison of presepsin concentration with serum for galactomannan (GM) and beta- D- glucan (BG) detection will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Káňová, MD,Ph.D., Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - Public Health Institute Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to make individual participant data available to other researchers.

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Masson S, Caironi P, Fanizza C, Thomae R, Bernasconi R, Noto A, Oggioni R, Pasetti GS, Romero M, Tognoni G, Latini R, Gattinoni L. Circulating presepsin (soluble CD14 subtype) as a marker of host response in patients with severe sepsis or septic shock: data from the multicenter, randomized ALBIOS trial. Intensive Care Med. 2015 Jan;41(1):12-20. doi: 10.1007/s00134-014-3514-2. Epub 2014 Oct 16. PMID 25319385
- [Background] Zhang J, Hu ZD, Song J, Shao J. Diagnostic Value of Presepsin for Sepsis: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2015 Nov;94(47):e2158. doi: 10.1097/MD.0000000000002158. PMID 26632748
- [Background] Ackland GL, Prowle JR. Presepsin: solving a soluble (CD14) problem in sepsis? Intensive Care Med. 2015 Feb;41(2):351-3. doi: 10.1007/s00134-014-3642-8. Epub 2015 Jan 22. No abstract available. PMID 25608923
- [Background] Okamura Y. [Usefulness of Presepsin Measurement: A New Biomarker for Sepsis]. Rinsho Byori. 2015 Jan;63(1):62-71. Japanese. PMID 26524880
- [Background] Rogic D, Juros GF, Petrik J, Vrancic AL. Advances and Pitfalls in Using Laboratory Biomarkers for the Diagnosis and Management of Sepsis. EJIFCC. 2017 May 1;28(2):114-121. eCollection 2017 May. PMID 28757819
- [Background] Endo S, Suzuki Y, Takahashi G, Shozushima T, Ishikura H, Murai A, Nishida T, Irie Y, Miura M, Iguchi H, Fukui Y, Tanaka K, Nojima T, Okamura Y. Usefulness of presepsin in the diagnosis of sepsis in a multicenter prospective study. J Infect Chemother. 2012 Dec;18(6):891-7. doi: 10.1007/s10156-012-0435-2. Epub 2012 Jun 13. PMID 22692596